CLINICAL TRIAL: NCT02140294
Title: Long Term Effect of Aggressive Nutritional Management on Survival in Patients With Alcoholic Liver Disease - A Randomized Control Trial
Brief Title: Long Term Effect of Aggressive Nutritional Management on Survival in Patients With Alcoholic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALD-01
Record Dates: First submitted 2014-04-09; First posted 2014-05-16 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polymeric nutritional supplement (Experimental)
  Interventions: Dietary Supplement: Polymeric nutritional supplements
- Standard Nutritional Treatment (Active Comparator)
  Interventions: Dietary Supplement: Standard Nutrional Treatment

INTERVENTIONS:
Dietary Supplement: Polymeric nutritional supplements
  Arms: Polymeric nutritional supplement
Dietary Supplement: Standard Nutrional Treatment
  Arms: Standard Nutritional Treatment

SUMMARY:
Patient found to be malnourished after the nutritional evaluation would be randomized in the two groups of the study. The control group would receive standard nutritional counseling from a trained dietician where as those in the intervention group would be given 120 gm of a polymeric nutritional supplement providing around 500 Kcal per day over and above the standard nutritional counseling from a trained dietician. Both the groups would receive standard medical treatment. The polymeric nutrient supplement would be taken by the patients in this arm for a period of 6 months.

DETAILED DESCRIPTION:
Patients with ALD (Alcoholic Liver Disease) would undergo a detailed clinical evaluation. Information would be collected regarding the onset and duration of symptoms, etiology, and severity of disease, other baseline clinical features, demographic characteristics, routine biochemical and hematological investigations, upper GI endoscopic findings and radiological investigations, patients would also be screened for the assessment of nutritional status. Patient found to be malnourished after the nutritional evaluation would be randomized in the two groups of the study. The control group would receive standard nutritional counseling from a trained dietician where as those in the intervention group would be given 120 gm of a polymeric nutritional supplement providing around 500 Kcal per day over and above the standard nutritional counseling from a trained dietician. Both the groups would receive standard medical treatment. The polymeric nutrient supplement would be taken by the patients in this arm for a period of 6 months. A record would be kept for the medications taken by the patients.

All the patients would be followed up at 1 week, 2 weeks, 3 weeks, 1 month, 2 months, 3 months, 6 months, and 1 year after inclusion. Clinical, nutritional and biological data were collected at each visit. All these patients would receive standard treatment of cirrhosis consisting of withdrawal from alcohol along with symptomatic treatment including B vitamins, diuretics, salt restriction, lactulose, beta blockers, and antibiotics after bacteriological samples if needed. All patients would receive endoscopic surveillance for portal hypertension. An adequate prophylaxis by ligation or beta blockers would be performed as needed. The patients with a past history of spontaneous bacterial peritonitis will receive antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive malnourished patients with ALD aged between 18 to 65 years of either gender would be enrolled.
* Abstinence of three months.

Exclusion Criteria:

* Severe alcoholic hepatitis
* Uncontrolled complication of the cirrhosis (variceal bleeding, infection, etc.),
* Hepatocellular carcinoma
* Ongoing corticosteroid treatment
* Co morbidities e.g. chronic renal insufficiency & Acquired immunodeficiency syndrome.
* Refusal to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess long term effect of aggressive nutritional management on survival. | 1 Year

SECONDARY OUTCOMES:
To assess long term effect of aggressive nutritional management on improvement in nutritional status. | 1 Year
  Nutritional Status will be measured by Royal Free Hospital-Global Assessment (RFH-GA) method.
To assess long term effect of aggressive nutritional management on onset or progression of complication. | 1 Year
To assess the effect of nutritional therapy on Health-related quality of life | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kalal C, Benjamin J, Shasthry V, Kumar G, Sharma MK, Joshi YK, Sarin SK. Effect of long-term aggressive nutrition therapy on survival in patients with alcohol-related cirrhosis: A randomized controlled trial. Indian J Gastroenterol. 2022 Feb;41(1):52-62. doi: 10.1007/s12664-021-01187-3. Epub 2022 Mar 2. PMID 35235198